CLINICAL TRIAL: NCT04630548
Title: The Safety and Efficacy of Immediate Post Placental IUD Insertion Versus the Post Puerperal IUD Insertion in Patients Undergoing Cesarean Delivery
Brief Title: Safety and Efficacy of Immediate Post Placental IUD Insertion in Patients Undergoing Cesarean Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moutaz Sherbini, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1401172
Record Dates: First submitted 2020-11-07; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: IUD
Keywords: IUD insertion; post placental insertion; puerperal insertion; cesarean section
MeSH Terms: interventions — Intrauterine Devices, Copper

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- post placental IUD insertion (Active Comparator): Following placental delivery, uterine cavity will be examined to exclude the presence of malformations or fibroids. Uterus will be stabilized by grasping it at fundus and the copper IUD (CuT 380 IUD) will be placed (within 10 minutes following the placental delivery) through the uterine wall incision high up in the uterine fundus (either by hand or using its applicator).
  Interventions: Device: Intrauterine copper device
- post puerperal IUD insertion (Active Comparator): IUD will be inserted 6 - 8 weeks following caesarean delivery (during the post puerperal visit).
  Interventions: Device: Intrauterine copper device

INTERVENTIONS:
Device: Intrauterine copper device — The obstetrical team will identify subjects who present in labor who meet the criteria and express interest in intrauterine contraception. Immediately after cesarean delivery, consented subjects will be randomized to immediate post placental IUD placement within 10 minutes or IUD placement at their routine standard postpartum visit (6 to 8 weeks postpartum).

SUMMARY:
Sixty six women who plan to deliver a live birth singleton via cesarean delivery who desire a Copper IUD for postpartum contraception will be approached for study participation thenvwill be randomized equally into two groups using computer generated numbers.

Group (A): (n=33) women IUD insertion post placental delivery (within 10mins) Group (B): (n=33) women IUD insertion post puerperal ( 6 to 8 weeks postpartum). Primary outcome will include IUD expulsion rate in both groups. Secondary outcomes will include other complications rates: missed threads (not seen by speculum examination), displaced IUD (more than 2 cm from the fundus in ultrasound), heavy puerperal bleeding, abdominal discomfort), Pregnancy rate, Discontinuation of the IUD usage and Satisfaction rate.

DETAILED DESCRIPTION:
Full history taking including a detailed history including medical and obstetric history, full obstetric examination and ultrasound evaluation to confirm gestational age and to exclude any of the exclusion criteria. Women who plan to deliver a live birth singleton via cesarean delivery at Kasr El-Ainy teaching will be considered for inclusion in the study. Women who desire a Copper IUD for postpartum contraception will be approached for study participation. The postpartum contraception plan will be documented during their prenatal course. It is also addressed by the obstetrical team upon admission to Labor & Delivery at El-Kasr El-Ainy teaching hospital. The obstetrical team will identify subjects who present in labor who meet the criteria and express interest in intrauterine contraception. Immediately after cesarean delivery, consented subjects will be randomized to immediate post placental IUD placement within 10 minutes or IUD placement at their routine standard postpartum visit (6 to 8 weeks postpartum).

For women randomized to the immediate post placental IUD insertion (n=33) the following will be done:

* after placental delivery, uterine cavity will be examined to exclude the presence of malformations or fibroids.
* Uterus will be stabilized by grasping it at fundus and the copper IUD (CuT 380 PREGNA IUD) will be placed (within 10 minutes following the placental delivery) through the uterine wall incision high up in the uterine fundus (either by hand or using its applicator).
* Before closing the uterine incision, the IUD strings will be guided to the lower uterine segment without trimming (If the cervix is closed, it should be dilated from above using a dilator).
* Enough care should be taken not to dislodge the IUD from its fundal position or to include the strings in uterine sutures.
* The IUD threads will protrude through the cervix in some cases its trimming will be done during follow-up if the patient is feeling any discomfort.
* Before discharge, the patient will be given a card including the intervention done (date & procedure), the follow-up schedule and investigator contacts. Also, they will be informed about normal postpartum symptoms, IUD side effects & possible complications (abdominal cramps, heavy puerperal bleeding, expulsion or protrusion of string) and instruct to seek medical help (to call the principle investigator) if any of the following warning signs have happened (severe lower abdominal pain, severe vaginal bleeding, infected discharge or lochia, fever, IUD expulsion & suspicion of pregnancy).

Subjects who are randomized for IUD insertion at their post puerperal visit will be assisted in scheduling a postpartum visit and IUD placement with their usual obstetrical care provider.

For women randomized for IUD insertion at their postpartum visit (n=33) the following will be done:(n=33):

* IUD will be inserted 6 - 8 weeks following caesarean delivery (during the post puerperal visit).
* Vaginal speculum will be inserted to expose the cervix & to exclude concomitant infection or bleeding.
* The anterior lip of the cervix will be grasped using ring forceps followed by uterine sounding to assess uterine cavity length.
* The IUD loaded sheath applicator (CuT 380 PREGNA IUD) will be introduced gently through the cervical canal and advanced slowly towards the uterine fundus.
* When fundal placement is confirmed, IUD will be released & the sheath will be withdrawn followed by trimming of the IUD string at 1 cm below the level of cervix.
* Following the insertion, transvaginal ultrasound (TVUS) will be done to assure fundal placement.
* Difficulties in insertion and patient discomfort will be recorded. Before leaving the clinic, the patient will be given a card including the intervention done (date & procedure), the follow-up schedule and investigator contacts. Also, they will be informed about potential IUD side effects & possible complications (abdominal cramps, vaginal bleeding, expulsion) and instruct to seek medical help (to call the principle investigator) if any of the following warning signs have happened (severe lower abdominal pain, severe vaginal bleeding, infected discharge, fever, IUD expulsion & suspicion of pregnancy).

All women who are going to have their IUD placement in post puerperal visits their contact numbers will be taken.

follow-up visits at 6 weeks ,3 & 6 months post-insertion will be scheduled. At 6 weeks post-insertion visit, participants (will be assessed via ultrasound and (to detect IUD expulsion or displacement) and speculum examination ( to detect presence of IUD threads).

At 3 months post-insertion visit, all subjects will be examined. Examination will include ultrasound (to detect IUD expulsion or displacement) and speculum examination ( to detect presence of IUD threads if not detected at 6 weeks post-insertion visit).

At 6 months post-insertion visit, all subjects will be examined & answering a simple questionnaire. Examination will include ultrasound (to detect IUD expulsion or displacement) and speculum examination ( to detect presence of IUD threads if not detected at 3 months post-insertion visit). The questionnaire will include questions regarding they have had a known expulsion, pregnancy event, or elective IUD removal and about the ease of placement and overall satisfaction with the timing of placement.

ELIGIBILITY:
Inclusion Criteria:

* Singleton full term pregnancy at ≥37 weeks gestation confirmed by LMP and first trimesteric ultrasound.
* Desired copper IUD placement for postpartum contraception.
* Candidate for cesarean delivery.
* Regional anesthesia.

Exclusion Criteria:

* Anatomic uterine abnormalities distorting the uterine cavity (obstructive myomata, bicornuate, septate, etc)
* Chorioamnionitis (also consider other risk factors such as prolonged rupture of membranes >18 hours, prolonged labor >24 hours, fever >38C).
* Puerperal sepsis.
* Unresolved postpartum hemorrhage.
* Known or suspected untreated endocervical gonorrhea, chlamydia.
* Wilson's disease, copper allergy (Paragard only).
* Known or suspected cervical or endometrial cancer or pelvic tuberculosis.
* Prolonged procedure > 2 hours.
* Preoperative hemoglobin 9.5 gm/dl.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
IUD expulsion rate | 6 months (following the insertion)
  to measure the frequency of IUD expulsion (IUD not found in ultrasound) following insertion by ultrasound examination.

SECONDARY OUTCOMES:
Missed threads rate (threads not seen by speculum examination) | 6 months (following the insertion)
  to measure the frequency of absent threads (threads not seen by speculum examination) following insertion.
displaced IUD rate | 6 months (following the insertion)
  to measure the frequency of displaced IUD (IUD more than 2 cm from the uterine fundus in ultrasound) following insertion.
pregnancy rate | within the 1st 6 months after insertion
  occurrence of any pregnancy event
satisfaction rate | 6 months after insertion
  by using questionnaire that include questions regarding they have had a known expulsion, pregnancy event, or elective IUD removal and about the ease of placement and overall satisfaction with the timing of placement.

CONTACTS AND LOCATIONS:
Overall Officials: moutaz M ELsherbini, MD, Principal Investigator — assistant professor (faculty of medicine -Cairo University

IPD SHARING:
Plan to Share IPD: No